CLINICAL TRIAL: NCT03181568
Title: A 12-week, Single-blind, Prospective, Randomized, Controlled, Pilot Clinical Trial to Evaluate Surface Area Reduction With Use of the MolecuLight i:X™ Imaging Device Compared to Standard Treatment of Chronic Wounds
Brief Title: Evaluating Surface Area Reduction Using MolecuLight Imaging Device
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Calver Pang (Other Government)
Responsible Party: Sponsor-Investigator, Calver Pang, Dr, Bradford Teaching Hospitals NHS Foundation Trust
Organization: Bradford Teaching Hospitals NHS Foundation Trust (Other Government)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: BTHFT 2159
Record Dates: First submitted 2017-06-06; First posted 2017-06-09 (Actual); Last update posted 2017-06-09 (Actual); Status verified 2017-06

CONDITIONS: Wound; Wound Infection
MeSH Terms: conditions — Wounds and Injuries; Wound Infection

STUDY DESIGN:
Intervention Model Description: This will be a single blinded randomised trial where the control group will be receiving a standard wound care whereas the treatment group would also be receiving standard wound care but under the guidance of the imaging device.
Who Masked: Care Provider, Investigator
Masking Description: Investigator will be blinded to study Clinical staff that will evaluate wounds at baseline, 2, 4, 6, 8, 10 and 12 weeks after date of randomisation and therapy initiation will be blinded
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (Other): This arm group (control) will receive standard wound care of chronic wounds
  Interventions: Procedure: Wound care
- Treatment (Other): The treatment arm of the study will utilize the MolecuLight i:X Imaging Device to guide a clinician to inspect, sample, debride or further evaluate areas within or around a wound where fluorescent bacteria are present
  Interventions: Device: MolecuLight i:X™ Imaging Device

INTERVENTIONS:
Device: MolecuLight i:X™ Imaging Device — Offers real-time detection of important biological and molecular information of a wound. The MolecuLight i:X Imaging Device is intended to assist clinicians during care and management of patients with chronic wounds by screening for the presence of potentially harmful bacteria levels. The device can capture and document either an image or video of the wound where the presence of fluorescent bacteria appears under violet light illumination. This information can be used to guide a clinician to inspect, sample, debride or further evaluate areas within or around a wound where fluorescent bacteria are present.
  Arms: Treatment
Procedure: Wound care — Standard wound care of chronic wounds e.g. sampling, debridement, infection control
  Arms: Control

SUMMARY:
12-week single-blind, prospective, randomized, controlled, pilot clinical trial assessing The MolecuLight i:X Imaging Device in chronic wounds. This device guides clinicians to inspect, sample, debride or further evaluate areas within or around a wound where potentially harmful bacteria appear under violet light illumination resulting in better overall care and accelerated surface area reduction compared to current standard care. The study aims to determine if this device aids in the healing of chronic wounds by reduction in size of wound compared to current standard of care.

DETAILED DESCRIPTION:
This is a prospective, 12-week, single-blinded, randomized, controlled clinical trial has been designed with two primary objectives needed to inform more comprehensive studies at a later date. We propose to evaluate the following two primary outcomes: (1) the ability of the MolecuLight i:X Imaging Device to predict non healing wounds and wounds at risk or infection (control arm) and (2) whether utilization of the MolecuLight i:X Imaging Device in guiding clinicians to inspect, sample, debride or further evaluate areas within or around a wound where fluorescent bacteria are present (treatment arm) increases wound healing rates relative to standard care (control arm) for the treatment of chronic wounds.

Both arms will receive standard procedures associated with wound care (e.g., sampling, debridement, preventative care, infection control, etc.) according to best practice guidelines. Patients will be randomly assigned to either the control or treatment arm and be followed as per the study protocol every time their wound is cared for over a 12-week period. The effectiveness of the MolecuLight i:X Imaging Device will be assessed with evaluation of wound surface area reduction rate and infection rates (incidence of infection and time to eradicate infection) compared to standard care.

All subjects randomized will be evaluated for 12 weeks from the date of enrollment and treatment initiation. Subjects who may have wound closure within the 12-week study period will continue to have scheduled study evaluation visits up to the end of week 12.

ELIGIBILITY:
Inclusion Criteria:

1. age ≥ 18 years
2. having a chronic wound that is not a diabetic foot ulcer
3. presence of the wound for ≥ 6 weeks and ≤ 2 years.
4. wound size surface area ≥ 2 cm2 and ≤ 50 cm2.
5. Willingness to comply with prescribed wound care regimen

Exclusion Criteria:

1. candidate for surgery in the next 12 weeks
2. a wound with necrotic tissue unable to tolerate debridement
3. uncontrolled diabetics (defined as HbA1c of >85.5mmol/mol)
4. presence of a diabetic foot ulcer
5. currently taking medication that may interfere with wound healing (e.g., oral systemic steroids, immunosuppressive drugs, unfractionated heparin infusion)
6. women who are currently pregnant or are breast feeding; or women of child bearing potential who are not currently taking adequate birth control
7. participation in another investigative drug or device trial currently or within the last 30 days

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2017-07-10 (Estimated); Primary Completion 2017-09-29 (Estimated); Study Completion 2017-09-29 (Estimated)

PRIMARY OUTCOMES:
Change in wound measurements at various time-points through the study | At baseline, 2nd, 4th, 6th, 8th, 10th and 12th week of the study
  These measurements will be made using the MolecuLight quickSize measurement tool, which will be loaded onto the i:X device. Wound measurements will be made after any wound cleaning and/or debridement, as per standard practice.
Change in wound characteristics at various time-points through the study | at baseline, 2, 4, 6, 8, 10 and 12 weeks
  Wound characteristics will be noted using the Bates-Jensen Wound Assessment score tool

CONTACTS AND LOCATIONS:
Locations (1):
- Bradford Teaching Hospitals NHS Trust, Bradford, United Kingdom

IPD SHARING:
Plan to Share IPD: No